CLINICAL TRIAL: NCT03256838
Title: A Long-Term, Open-Label, Prospective Phase IV Study to Assess the Safety and Efficacy of Nephoxil® in Subjects With End Stage Renal Disease (ESRD) on Dialysis
Brief Title: Assess the Safety and Efficacy of Nephoxil® in Subjects With End Stage Renal Disease (ESRD) on Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBB00501
Record Dates: First submitted 2017-07-24; First posted 2017-08-22 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Kidney Failure, Chronic; End-stage Renal Disease; Phosphorus Metabolism Disorders; Hyperphosphatemia
Keywords: Citric Acid; Ferric Compounds; Renal Insufficiency; Anticoagulants; Calcium Chelating Agents; Chelating Agents; Sequestering Agents; Hemodialysis; Dialysis; Renal Failure; Kidney Failure; Urologic Diseases; Metabolic Disease; Kidney Diseases; Renal Insufficiency, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Phosphorus Metabolism Disorders; Hyperphosphatemia; Renal Insufficiency; Urologic Diseases; Metabolic Diseases; Kidney Diseases; Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric citrate (Experimental): Ferric Citrate (Nephoxil® Capsules) will be dosed three times a day (with meals).
  Interventions: Drug: Ferric Citrate

INTERVENTIONS:
Drug: Ferric Citrate — Ferric citrate will be provided as a 500mg capsule. All intervention doses will be based on serum phosphorus levels.
  Other Names: Nephoxil® Capsules

SUMMARY:
To assess the long-term safety and effectiveness of Nephoxil® for the treatment of hyperphosphatemia in patients with ESRD undergoing dialysis.

DETAILED DESCRIPTION:
This study is an open-label, prospective, long term, Phase IV study to assess the safety and efficacy of Nephoxil® in subjects with ESRD on dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≧ 18 years of age on the day of signing informed consent or other age required by local regulation
2. Willing and able to provide written informed consent
3. ESRD patients who is undergoing hemodialysis 3 times per week and is considered necessary to receive medication for hyperphosphatemia by his/her treating physician
4. Serum ferritin <1000 ng/mL and transferrin saturation (TSAT) < 50% at the Enrollment Visit
5. Women of child-bearing potential (WOCBP [defined as women ≤ 50 years of age with a history of amenorrhea for < 12 months prior to study entry]) who is willing to use an effective form of contraception during study participation

Exclusion Criteria:

1. Has any known contraindication to ferric citrate according to locally approved prescribing information, include but not limited to the following criteria:

   i. Is allergic to ferric citrate ii. Has hypophosphatemia iii. Has hemochromatosis or iron overload syndromes iv. Has active severe GI disorders
2. Has parathyroidectomy (PTx) or percutaneous ethanol injection therapy (PEIT) within 3 months prior to Enrollment Visit or serum calcium < 7 mg/dL at the Enrollment Visit
3. Has participated in another interventional study for any investigational agent or device within 30 days prior to enrollment
4. Is currently pregnant or breastfeeding
5. Other unstable medical condition or psychiatric conditions that is considered unsuitable for this study per Investigator's clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | 13 months
  Number of subjects with treatment-emergent adverse events (TEAEs)
Percentage of subjects with treatment-emergent adverse events (TEAEs) | 13 months
  Percentage of subjects with treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Serum Phosphorus | 13 months
  Serum Phosphorus will be assessed by time-course changes of serum phosphorus levels and proportion of subjects achieved target range of serum phosphorus (>=3.5 mg/dL and <=5.5. mg/dL) from baseline to the end-of-treatment.

OTHER OUTCOMES:
Serum calcium | 13 months
  Time-course changes of serum calcium from baseline.
Intact plasma parathyroid hormone (iPTH) | 13 months
  Time-course changes of intact plasma parathyroid hormone (iPTH) from baseline.
Ferritin | 13 months
  Time-course changes of ferritin from baseline.
Transferring saturation (TSAT) percentage | 13 months
  Time-course changes of transferring saturation (TSAT) percentage from baseline.
Serum iron | 13 months
  Time-course changes of serum iron from baseline.
Total iron-binding capacity (TIBC) | 13 months
  Time-course changes of total iron-binding capacity (TIBC) from baseline.
Hemoglobin | 13 months
  Time-course changes of hemoglobin from baseline.
Dose of IV iron | 13 months
  Time-course changes of dose of IV iron from baseline.
Dose of erythropoiesis stimulating agents (ESA) | 13 months
  Time-course changes of dose of erythropoiesis stimulating agents (ESA) from baseline.
Treatment adherence | 13 months
  Prescribed dose and the dose actually taken at each time point will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Szu Wu, M.D., Principal Investigator — Division of Nephrology, Department of Internal Medicine, Taipei Medical University Hospital
Locations (9):
- Taiwan (9):
  - Division of Nephrology, Department of Internal Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Division of Nephrology, Department of Internal Medicine, Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City
  - Division of Nephrology, Department of Internal Medicine, Keelung Chang Gung Memorial Hospital, Keelung
  - Division of Nephrology, Department of Internal Medicine, Far East Memorial Hospital, New Taipei City
  - Division of Nephrology, Department of Internal Medicine, Taichung Veterans General Hospital, Taichung
  - Division of Nephrology, Department of Internal Medicine, National Taiwan University Hospital, Taipei
  - Division of Nephrology, Department of Internal Medicine, Taipei Medical University Hospital, Taipei
  - Division of Nephrology, Department of Internal Medicine, Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Division of Nephrology, Department of Internal Medicine, Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CT, Lee CC, Wu MJ, Chiu YW, Leu JG, Wu MS, Peng YS, Wu MS, Tarng DC. Long-term safety and efficacy of ferric citrate in phosphate-lowering and iron-repletion effects among patients with on hemodialysis: A multicenter, open-label, Phase IV trial. PLoS One. 2022 Mar 3;17(3):e0264727. doi: 10.1371/journal.pone.0264727. eCollection 2022. PMID 35239732